CLINICAL TRIAL: NCT04446481
Title: Tuning Up Memory-related Brain Potentials Using Real-time Neurofeedback in Older Veterans
Brief Title: Neurofeedback to Aid Vets' Memory
Acronym: TUNe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N3173-P; RX-003173 (Other Grant/Funding Number: Department of Veterans Affairs); JIA-20-003-HE (Other: VA IRB)
Record Dates: First submitted 2020-06-03; First posted 2020-06-25 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Impairment
Keywords: neurofeedback; amnestic MCI; wireless EEG; Bluegrass Memory Test; working memory
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Neurofeedback; Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: Exp1. Protocol establishment: 15 cognitively intact and 15 Vets with mild cognitive impairment
  Exp2. Efficacy Testing: 20 Vets over the age of 60
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MCI patients (Experimental): Vets with mild cognitive impairment
  Interventions: Device: Neurofeedback
- NC (Active Comparator): Normal healthy Veterans
  Interventions: Device: Neurofeedback

INTERVENTIONS:
Device: Neurofeedback — Neurofeedback will be tested in both groups of Vets
  Other Names: biofeedback

SUMMARY:
Military deployment is associated with increased risk of mild cognitive impairment (MCI). Combat stress related memory deficits has been well documented. Mild cognitive impairment such as memory deficits are the most common and earliest symptoms of Alzheimer's disease and related dementia (ADRD). The complaints about declined memory are common in healthy and cognitively intact civilian older adults, but less understood in aging Veterans. Brain training strategies to enhance cognitive skills and especially memory processes are unmet needs in aging Veterans who are at additional risk for MCI induced by ADRD. Since currently there is no effective drug treatment to stop cognitive decline, non-invasive brain training to boost memory functions in older Veterans is an increasingly attractive option to attenuating decline in memory.

DETAILED DESCRIPTION:
The proposed project is poised to investigate state-of-art neurofeedback (NF; biofeedback of brain activity) training for self-modulation of neural plasticity to boost memory performance in Veterans. The recent advance of NF with Brian-Computer Interface (BCI) has provided a novel way to examine brain functions and plasticity. Thus far, there have been limited applications that have developed effective experimental and clinical paradigms for rehabilitation in Veterans. Historically, brainwave patterns during memory task performance have been analysed offline, a methodology which does not allow real-time NF modulation and training. The central hypothesis guiding this research is that optimal memory-related brainwave patterns of a Veteran can be trained. The online NF allows maximization of brainwave patterns associated with healthier memory states.

The development of efficient NF paradigms to augment memory performance is an important first step for the application of this nonpharmacologic intervention to improve combat Veterans' memory functions and potential for treating MCI due to mild TBI or pain. The pilot work will start with wider range of Veterans using state-of-the-art wearable wireless brain-computer interface headset, which is affordable and can be easily set up in VAMCs and eventually in remote assessment settings. This innovative, cognitive neuroscience based, nonpharmacologic intervention serves to revolutionize the diagnosis and treatment of combat Veterans who are at risk for degenerative dementia.

ELIGIBILITY:
Inclusion Criteria:

* Veterans age 60 and older

Exclusion Criteria:

* Veterans diagnosed with PTSD, epilepsy schizophrenia, or use benzodiazepines

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
EEG alpha band | 6-8 weeks
  alpha power under eyes closed and eyes open are linked to better mental state; likely biomarker for mild cognitive impairment.

SECONDARY OUTCOMES:
memory-related potentials | 6-8 weeks
  Brainwaves that are linked to better memory performance
California Verbal Learning Test | About 6-8 weeks
  A battery of neuropsychological testing cognitive functions

CONTACTS AND LOCATIONS:
Overall Officials: Yang Jiang, PhD, Principal Investigator — Lexington VA Medical Center, Lexington, KY
Locations (1):
- Lexington VA Medical Center, Lexington, KY, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be analyzed and kept at least 6 years after project. Results will be shared via publications. The qualified researchers may contact PI and VA for further sharing of the research data.

REFERENCES:
- [Result] Jiang Y, Jessee W, Hoyng S, Borhani S, Liu Z, Zhao X, Price LK, High W, Suhl J, Cerel-Suhl S. Sharpening Working Memory With Real-Time Electrophysiological Brain Signals: Which Neurofeedback Paradigms Work? Front Aging Neurosci. 2022 Mar 28;14:780817. doi: 10.3389/fnagi.2022.780817. eCollection 2022. PMID 35418848
- [Result] Jiang Y, Neal J, Sompol P, Yener G, Arakaki X, Norris CM, Farina FR, Ibanez A, Lopez S, Al-Ezzi A, Kavcic V, Guntekin B, Babiloni C, Hajos M. Parallel electrophysiological abnormalities due to COVID-19 infection and to Alzheimer's disease and related dementia. Alzheimers Dement. 2024 Oct;20(10):7296-7319. doi: 10.1002/alz.14089. Epub 2024 Aug 29. PMID 39206795
- See also: Sharpening Working Memory With Real-Time Electrophysiological Brain Signals: Which Neurofeedback Paradigms Work? — https://www.frontiersin.org/journals/aging-neuroscience/articles/10.3389/fnagi.2022.780817/full

DOCUMENTS (1):
  • Informed Consent Form (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/81/NCT04446481/ICF_000.pdf